CLINICAL TRIAL: NCT02748512
Title: A Controlled, Multi-Center Study of the Utilization and Safety of the MkII Inserter and the Safety of the FAI Insert in Subjects With Non-Infectious Uveitis Affecting the Posterior Segment of the Eye.
Brief Title: Utilization and Safety of the Mk II Inserter and the Safety of the FAI Insert in Non-Infectious Uveitis
Acronym: MkII
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: EyePoint Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PSV-FAI-006
Record Dates: First submitted 2016-04-19; First posted 2016-04-22 (Estimated); Results first posted 2020-05-01 (Actual); Last update posted 2020-05-01 (Actual); Status verified 2020-04

CONDITIONS: Non-Infectious Uveitis
MeSH Terms: interventions — Fluocinolone Acetonide

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes

ARMS (2):
- FAI Insert administered using the Mk II inserter (Experimental): The test article is the Fluocinolone Acetonide Intravitreal (FAI) insert, which contains 0.18 mg FA and delivers FA into the vitreous humor for 36 months, at a nominal rate of approximately 0.2 μg FA/day. The FAI insert will be administered to the study eye as an intravitreal injection through the pars plana.
  Interventions: Drug: FAI Insert administered using the Mk II inserter
- FAI Insert administered using the Mk I inserter (Active Comparator): The test article is the Fluocinolone Acetonide Intravitreal (FAI) insert, which contains 0.18 mg FA and delivers FA into the vitreous humor for 36 months, at a nominal rate of approximately 0.2 μg FA/day. The FAI insert will be administered to the study eye as an intravitreal injection through the pars plana.
  Interventions: Drug: FAI Insert administered using the Mk I inserter

INTERVENTIONS:
Drug: FAI Insert administered using the Mk II inserter
  Other Names: Fluocinolone Acetonide Intravitreal (FAI)
  Arms: FAI Insert administered using the Mk II inserter
Drug: FAI Insert administered using the Mk I inserter
  Other Names: Fluocinolone Acetonide Intravitreal (FAI)
  Arms: FAI Insert administered using the Mk I inserter

SUMMARY:
This trial is a 12 month, Phase 3, multi-center, randomized, single-masked (subject), controlled study designed to evaluate the utilization and safety of the Mk II inserter and the safety of the FAI insert, in subjects with non-infectious uveitis affecting the posterior segment of the eye.

DETAILED DESCRIPTION:
This trial is a 12 month, Phase 3, multi-center, randomized, single-masked (subject), controlled study designed to evaluate the utilization and safety of the MK II inserter and the safety of the FAI insert, in subjects with non-infectious uveitis affecting the posterior segment of the eye.

ELIGIBILITY:
Inclusion Criteria:

1. Male or non-pregnant female at least 18 years of age at time of consent
2. At least one eye has a history of non-infectious uveitis affecting the posterior segment
3. Subject has ability to understand and sign the Informed Consent Form
4. Subject is willing and able to comply with study requirements

Exclusion Criteria:

1. Allergy to fluocinolone acetonide or any component of the FAI insert
2. Ocular malignancy in either eye, including choroidal melanoma
3. Uveitis with infectious etiology
4. Current viral diseases of the cornea and conjunctiva including epithelial herpes simplex keratitis (dendritic keratitis), vaccinia, and varicella
5. Current mycobacterial infections of the eye or fungal diseases of ocular structures
6. Subjects who yield, during screening, a confirmed positive test for human immune deficiency virus (HIV) or syphilis
7. Systemic infection within 30 days prior to study Day 1
8. Peripheral retinal detachment in area of insertion
9. Elevated intraocular pressure (IOP) > 21 mmHg, or chronic hypotony < 6 mmHg
10. Concurrent therapy at screening with IOP-lowering pharmacologic agent in the study eye
11. Current diagnosis of any form of glaucoma or ocular hypertension in study eye at Screening, unless study eye has been previously treated with an incisional surgery procedure that has resulted in stable IOP in the normal range (10-21 mmHg)
12. Known history of clinically significant IOP elevation in response to steroid treatment in either eye, unless study eye has been previously treated with an incisional surgery procedure that has resulted in stable IOP in the normal range (10-21 mmHg)
13. Ocular surgery or capsulotomy performed on the study eye within 30 days prior to study Day 1
14. Intravitreal treatment of study eye: with FAI insert within 36 months prior to study Day 1;with Retisert within 30 months prior to study Day 1; with Ozurdex within 90 days prior to study Day 1; or with Triesence or Trivaris within 30 days prior to study Day 1
15. Peri-ocular or subtenon steroid treatment of study eye within 30 days prior to study Day 1
16. Treatment with an investigational drug or device within 30 days prior to study Day 1, except the FAI insert within this protocol
17. Pregnant or nursing females; females of childbearing potential who are unwilling or unable to use an acceptable method of contraception as outlined in this protocol from at least 14 days prior to study Day 1 until the Month 12 Visit
18. Any condition which, in the judgment of the Investigator, could make the subject inappropriate for entry into this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2016-02-23 (Actual); Primary Completion 2017-08-17 (Actual); Study Completion 2017-08-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Flavio Leonin Jr., MD, Principal Investigator — pSivida Corp, Senior Manager, Clinical Affairs; Gerard E Riedel, PhD, Study Chair — pSivida Corp, Vice President, Regulatory Affairs; Paul Ashton, PhD, Study Director — pSivida Corp, Chief Executive Officer
Locations (6):
- United States (6):
  - Retina Consultants of Southern Colorado, PC, Colorado Springs, Colorado
  - Massachusetts Eye Research and Surgery Institution / Ocular Immunology & Uveitis Foundation, Waltham, Massachusetts
  - Duke Eye Center, Durham, North Carolina
  - Cleveland Clinic Foundation Cole Eye Institute, Cleveland, Ohio
  - Charleston Neuroscience Institute, Ladson, South Carolina
  - Texas Retina Associates, Arlington, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: One subject was assigned to the Mk II; however, received treatment with the Mk I after attempted to use 2 different Mk II inserters without success and switched to the Mk I inserter. The data for this subject were included in the Mk II inserter treatment group for ITT population and in the Mk I inserter treatment group for the safety population
Pre-assignment Details: Prior to analysis no Subjects were Excluded From the Utilization Analysis (i.e., completed Day 7). 1 MKI and 1 MKII eyes were lost to follow-up at Month 12.
Units Other Than Participants: Eyes
Groups:
- Mk II Inserter: Fluocinolone Acetonide Intravitreal (FAI) Insert, administered using the Mk II inserter
- Mk I Inserter: Fluocinolone Acetonide Intravitreal (FAI) Insert, administered using the Mk I inserter
Period: Overall Study
Arm/Group | Mk II Inserter | Mk I Inserter
Started | 14; 27 Eyes | 12; 11 Eyes
Completed (14 subjects had 1 study eye treated and 12 subjects had 2 study eyes treated) | 13; 26 Eyes | 11; 10 Eyes
Not Completed | 1; 1 Eyes | 1; 1 Eyes
Not completed — Lost to Follow-up | 1 | 1

BASELINE CHARACTERISTICS:
Units Other Than Participants: Eyes
Groups:
- FAI Insert Administered Using the Mk II Inserter: The test article is the Fluocinolone Acetonide Intravitreal (FAI) insert, which contains 0.18 mg FA and delivers FA into the vitreous humor for 36 months, at a nominal rate of approximately 0.2 μg FA/day. The FAI insert will be administered to the study eye as an intravitreal injection through the pars plana.
  FAI Insert administered using the Mk II inserter
- FAI Insert Administered Using the Mk I Inserter: The test article is the Fluocinolone Acetonide Intravitreal (FAI) insert, which contains 0.18 mg FA and delivers FA into the vitreous humor for 36 months, at a nominal rate of approximately 0.2 μg FA/day. The FAI insert will be administered to the study eye as an intravitreal injection through the pars plana.
  FAI Insert administered using the Mk I inserter
- Total: Total of all reporting groups
Arm/Group | FAI Insert Administered Using the Mk II Inserter | FAI Insert Administered Using the Mk I Inserter | Total
Number analyzed (Participants) | 14 | 12 | 26
Number analyzed (Eyes) | 27 | 11 | 38
Age, Continuous [Mean (Standard Deviation); unit: Years] | 51.3 (11.82) | 48.9 (11.19) | 50.4 (12.12)
Sex: Female, Male [Count of Units; unit: Eyes]
  Female | 18 | 7 | 25
  Male | 9 | 4 | 13
Race/Ethnicity, Customized [Count of Units; unit: Eyes]
  White | 21 | 8 | 29
  Black or African American | 5 | 3 | 8
  Asian | 1 | 0 | 1
Region of Enrollment [Number; unit: Eyes]
  United States | 27 | 11 | 38
Overall Eyes Evaluated [Count of Units; unit: Eyes] | 27 | 11 | 38

OUTCOME MEASURES:

1. Primary Outcome: The Utilization of the Mk II Inserter From the Day of Treatment Through 7 Days Following Treatment.
Description: The primary utilization endpoint was defined as the proportion of intravitreal insertion procedures that were assessed by the investigator as satisfactory. A satisfactory procedure was defined as one receiving a score from the Investigator as either Very Easy, Easy, or Routine.
Time Frame: Day 7
Population: Intent-to-treat population - Assessment Categories
Measure: Count of Units; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Mk II Inserter | Mk I Inserter
Number analyzed (Participants) | 14 | 12
Number analyzed (Eyes) | 27 | 11
Eyes
  Very Easy | 10 | 3
  Easy | 3 | 2
  Routine | 5 | 0
  Difficult | 7 | 4
  Very Difficult | 2 | 2

2. Secondary Outcome: The Safety of the FAI Insert During 12 Months Following Treatment Reported as Percentages.
Description: To assess the safety of the FAI insert during 12 months following treatment reported as percentages.
Time Frame: Month 12
Population: Overall Summary of Treatment-Emergent Ocular Adverse Events at Month 12 (Safety Population). Note 27/11 (ITT Population) and 26/12 (Safety Population).
Measure: Count of Units; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Mk II Inserter | Mk I Inserter
Number analyzed (Participants) | 14 | 12
Number analyzed (Eyes) | 26 | 12
Eyes
  TEAE | 12 | 7
  Serious TEAE | 1 | 1
  Treatment-related TEAE | 10 | 4
  Treatment-related serious TEAE | 0 | 0
  TEAE leading to FAI insert removal | 0 | 1
  TEAE leading to study discontinuation | 0 | 0
  AE leading to death | 0 | 0

ADVERSE EVENTS:
Time Frame: Overall Summary of Treatment-Emergent Non-ocular and Ocular Adverse Events at Month 12 (Safety Population - MKII 26 eyes; MKI 12 eyes)
Description: Overall Summary of Treatment-Emergent Non-ocular and Ocular Adverse Events at Month 12 (Safety Population - MKII 26 eyes; MKI 12 eyes)
Arm/Group | Mk II Inserter | Mk I Inserter
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/12
Serious Adverse Events (participants affected / at risk) | 4/14 | 3/12
Other Adverse Events (participants affected / at risk) | 14/14 | 11/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Mk II Inserter (N=14) | Mk I Inserter (N=12)
Tachycardia (Cardiac disorders) | 1 | 1 — By-treatment counts were per treated eye and a subject could be included more than once. Total subject counts were per subject and a subject was included only once even if the subject had both eyes treated.
Pancreatitis (Gastrointestinal disorders) | 1 | 1 — By-treatment counts were per treated eye and a subject could be included more than once. Total subject counts were per subject and a subject was included only once even if the subject had both eyes treated.
Type 2 Diabetes Mellitus (Metabolism and nutrition disorders) | 1 | 1 — By-treatment counts were per treated eye and a subject could be included more than once. Total subject counts were per subject and a subject was included only once even if the subject had both eyes treated.
Renal Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 — By-treatment counts were per treated eye and a subject could be included more than once. Total subject counts were per subject and a subject was included only once even if the subject had both eyes treated.
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 1 — By-treatment counts were per treated eye and a subject could be included more than once. Total subject counts were per subject and a subject was included only once even if the subject had both eyes treated.
Retinal Detachment (Eye disorders) | 0 | 1
Factitious Disorder (Psychiatric disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Mk II Inserter (N=14) | Mk I Inserter (N=12)
Bronchitis (Infections and infestations) | 1 | 0 — By-treatment counts were per treated eye and a subject could be included more than once. Total subject counts were per subject and a subject was included only once even if the subject had both eyes treated.
Candida Infection (Infections and infestations) | 1 | 1 — By-treatment counts were per treated eye and a subject could be included more than once. Total subject counts were per subject and a subject was included only once even if the subject had both eyes treated.
Cellulitis (Infections and infestations) | 0 | 1 — By-treatment counts were per treated eye and a subject could be included more than once. Total subject counts were per subject and a subject was included only once even if the subject had both eyes treated.
Nasopharyngitis (Infections and infestations) | 1 | 0 — By-treatment counts were per treated eye and a subject could be included more than once. Total subject counts were per subject and a subject was included only once even if the subject had both eyes treated.
Oral Herpes (Infections and infestations) | 1 | 0 — By-treatment counts were per treated eye and a subject could be included more than once. Total subject counts were per subject and a subject was included only once even if the subject had both eyes treated.
Tooth Infection (Infections and infestations) | 0 | 1 — By-treatment counts were per treated eye and a subject could be included more than once. Total subject counts were per subject and a subject was included only once even if the subject had both eyes treated.
Urinary Tract Infection (Infections and infestations) | 1 | 0 — By-treatment counts were per treated eye and a subject could be included more than once. Total subject counts were per subject and a subject was included only once even if the subject had both eyes treated.
Diarrhoea (Gastrointestinal disorders) | 1 | 1 — By-treatment counts were per treated eye and a subject could be included more than once. Total subject counts were per subject and a subject was included only once even if the subject had both eyes treated.
Pancreatic cyst (Gastrointestinal disorders) | 1 | 0 — By-treatment counts were per treated eye and a subject could be included more than once. Total subject counts were per subject and a subject was included only once even if the subject had both eyes treated.
Toothache (Gastrointestinal disorders) | 0 | 1 — By-treatment counts were per treated eye and a subject could be included more than once. Total subject counts were per subject and a subject was included only once even if the subject had both eyes treated.
Gout (Metabolism and nutrition disorders) | 1 | 0 — By-treatment counts were per treated eye and a subject could be included more than once. Total subject counts were per subject and a subject was included only once even if the subject had both eyes treated.
Hypokalemia (Metabolism and nutrition disorders) | 1 | 1 — By-treatment counts were per treated eye and a subject could be included more than once. Total subject counts were per subject and a subject was included only once even if the subject had both eyes treated.
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 2 — By-treatment counts were per treated eye and a subject could be included more than once. Total subject counts were per subject and a subject was included only once even if the subject had both eyes treated.
Pituitary-dependent Cushing's syndrome (Endocrine disorders) | 1 | 1 — By-treatment counts were per treated eye and a subject could be included more than once. Total subject counts were per subject and a subject was included only once even if the subject had both eyes treated.
Laboratory test abnormal (Investigations) | 1 | 0 — By-treatment counts were per treated eye and a subject could be included more than once. Total subject counts were per subject and a subject was included only once even if the subject had both eyes treated.
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 — By-treatment counts were per treated eye and a subject could be included more than once. Total subject counts were per subject and a subject was included only once even if the subject had both eyes treated.
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 1 — By-treatment counts were per treated eye and a subject could be included more than once. Total subject counts were per subject and a subject was included only once even if the subject had both eyes treated.
Rash (Skin and subcutaneous tissue disorders) | 1 | 1 — By-treatment counts were per treated eye and a subject could be included more than once. Total subject counts were per subject and a subject was included only once even if the subject had both eyes treated.
Hypertension (Vascular disorders) | 2 | 0 — By-treatment counts were per treated eye and a subject could be included more than once. Total subject counts were per subject and a subject was included only once even if the subject had both eyes treated.
Anterior chamber cell (Eye disorders) | 0 | 1
Cataract (Eye disorders) | 4 | 1
Computer vision syndrome (Eye disorders) | 0 | 1
Conjunctival haemorrhage (Eye disorders) | 2 | 0
Eye pain (Eye disorders) | 0 | 1
Eye pruritus (Eye disorders) | 1 | 0
Lacrimation increased (Eye disorders) | 1 | 0
Macular fibrosis (Eye disorders) | 1 | 0
Meibomianitis (Eye disorders) | 1 | 0
Posterior capsule opacification (Eye disorders) | 1 | 0
Retinal detachment (Eye disorders) | 0 | 1
Retinal pigment epitheliopathy (Eye disorders) | 1 | 0
Retinal vascular disorder (Eye disorders) | 1 | 0
Subretinal fluid (Eye disorders) | 0 | 1
Uveitis (Eye disorders) | 1 | 0
Visual acuity reduced (Eye disorders) | 4 | 1
Vitreous haze (Eye disorders) | 1 | 0
Intraocular pressure decreased (Investigations) | 0 | 1
Intraocular pressure increased (Investigations) | 2 | 2
Device dislocation (Product Issues) | 1 | 1
Device failure (Product Issues) | 0 | 1
Injection site pain (General disorders) | 0 | 1
Factitious disorder (Psychiatric disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI is restricted from publicly releasing results.

DOCUMENTS (2):
  • Study Protocol (2016-04-04): https://cdn.clinicaltrials.gov/large-docs/12/NCT02748512/Prot_000.pdf
  • Statistical Analysis Plan (2016-04-12): https://cdn.clinicaltrials.gov/large-docs/12/NCT02748512/SAP_001.pdf